CLINICAL TRIAL: NCT00598884
Title: Internet-Based Self-Management Intervention for Prolonged Grief
Brief Title: Effectiveness of an Internet-Based Self-Management Program in Treating Prolonged Grief Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34MH079884 (NIH); R34MH079884 (NIH); DSIR 83-ATP
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Grief; Mental Health
Keywords: Clinical Protocols; Behavioral Research; Prevention
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 6-week delay start (Experimental): This group begins treatment 6 weeks after recruitment and baseline.
  Interventions: Behavioral: Internet-Based Self-Management for Prolonged Grief Symptoms
- No delay start (Experimental): This group begins treatment after enrollment and assessment with no wait period.
  Interventions: Behavioral: Internet-Based Self-Management for Prolonged Grief Symptoms

INTERVENTIONS:
Behavioral: Internet-Based Self-Management for Prolonged Grief Symptoms — The treatment consists of empirically derived cognitive behavioral therapy strategies to promote stable and active routines, self-care, accommodation of loss, enhanced self-efficacy, re-engagement in pleasurable activities, and reattachment with significant others. Treatment sessions will be Internet-based and will occur three times per week for 6 weeks.

SUMMARY:
This study will evaluate the effectiveness of an Internet-based self-help program in treating people who are at risk for developing prolonged grief disorder following a recent loss.

DETAILED DESCRIPTION:
Prolonged grief disorder (PGD) is a severe psychiatric condition that occurs in about 10% of people who experience a recent loss. PGD does not just go away with time and is associated with considerable functional impairment, physical and mental health problems, lost productivity, lack of interest in previously enjoyed activities, suicide, and depression. Because the majority of people with PGD are elderly and less capable of pursuing outside care, making readily available treatments for PGD is very important. Current treatments for PGD include psychotherapy and antidepressant medications, but there is very little solid research on the effectiveness of these treatments. Previous studies have shown that Internet-based mental health treatments are an effective and cost-efficient way to provide self-help to people who otherwise would not seek care. Using strategies from the psychotherapy known as cognitive behavioral therapy (CBT), this study will evaluate the effectiveness of an Internet-based self-help program in treating people who are at risk for developing prolonged grief disorder following a recent loss.

This is a randomized, wait-list control design. Participants will be randomized to immediately begin the intervention or to wait for 6-weeks before beginning. The intervention will ask participants to log-on to the study's self-help website three times per week for the 6 weeks of treatment. During these sessions, participants will be offered optional information about grief and coping with grief and will be required to complete computer exercises that involve identifying self-care needs, support systems, and short- and long-term goals. Participants will also be asked to perform off-line activities that are designed to increase self-care and social activities and that may take anywhere from a few minutes to 30 minutes per day. For all participants, there will be four assessments, after randomization, before beginning treatment (these 2 are the same for the immediate group), upon completion of the intervention, at 6 weeks post-intervention, at 3 months post-intervention (for immediate group). Assessments will include questions about mental and physical health adjustment, beliefs about the loss, and coping status.

ELIGIBILITY:
Inclusion criteria:

* Meets criteria for a diagnosis of prolonged grief (with the exception of the requirement for 6-month duration of symptoms) using the Prolonged Grief -13
* Access to the Internet

Exclusion Criteria:

* Lifetime history of bipolar disorder, schizophrenia, psychosis, or delusional disorders
* History of substance or alcohol dependence other than nicotine in the year prior to study entry
* Significant suicidal ideation
* Concurrent psychotherapy initiated within 3 months prior to study entry, or ongoing psychotherapy specifically targeting loss; general supportive therapy initiated more than 3 months prior to study entry is acceptable

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2009-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Prolonged grief symptoms and other comorbid mental health difficulties | Measured at Weeks pre-, post-, 6-week, 3-month

SECONDARY OUTCOMES:
Social functioning and coping styles | Measured at pre-, post-, 6-week, 3-month

CONTACTS AND LOCATIONS:
Overall Officials: Brett T. Litz, PhD, Principal Investigator — Boston University
Locations (1):
- Boston VA Medical Center, Boston, Massachusetts, United States